CLINICAL TRIAL: NCT03812315
Title: Antimicrobial Effect OF Propolis Administrated Through Two Different Vehicles In High Caries Risk Children: A Randomized Clinical Trial
Brief Title: Antimicrobial Effect OF Propolis Administrated Through Two Different Vehicles In High Caries Risk Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Clinical Instructor, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Propolis in 2 vehicles
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Early Childhood Caries
Keywords: Propoplis; chewing gum; mouthwash; high caries risk children; antimicrobial

STUDY DESIGN:
Intervention Model Description: The study is a two parallel arms randomized controlled clinical trial where 60 high caries risk children of 6-8 years will be selected from outpatient clinic of Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Alexandria University, after securing the necessary consents. The children will be divided randomly into two equal groups (30 children each)
Who Masked: Outcomes Assessor
Masking Description: The investigator and the participants will not be blinded to the treatment type as each group has to be given different instruction according to their treatment protocol. However, the statistician and the microbiologist will be blinded to the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propolis chewing gum (Experimental): 2 % pure raw propolis, 20-35% gum base, 2.5% flavors, 0.3% sorbitol and 0.3% coloring substance. Children will be instructed to chew the specially prepared propolis chewing gum for at least 20 minutes, twice daily, after breakfast and before bedtime.
  Interventions: Combination Product: Propolis chewing gum
- Propolis mouthwash (Active Comparator): The formulation includes 2% pure raw propolis, 40 ml flavors, 150 ml propylene glycol, 60 gm sorbitol, 0.1 g coloring substance and water. Children will be instructed to rinse using the prepared propolis mouthwash for 1 min, twice a day, after breakfast and before bedtime.
  Interventions: Combination Product: Propolis mouthwash

INTERVENTIONS:
Combination Product: Propolis chewing gum — Children who will use chewing gum will be instructed to chew a gum for 20 minutes once after breakfast and another before bed time for two weeks.
  Arms: Propolis chewing gum
Combination Product: Propolis mouthwash — Children who will use mouthwash will be instructed to rinse with 10 ml for 60 seconds twice daily once after breakfast and another before bedtime for two weeks.
  Arms: Propolis mouthwash

SUMMARY:
Propolis is a natural product collected by bees to seal holes and repair structures in their hives. Recently it has attracted much attention as useful substance applied in medicine and cosmetics thanks to its antimicrobial properties. Contemporary dentistry is an inseparable part of medicine and therefore attempts were made to use propolis in dentistry, as well.

Purpose of the study: to investigate the effect of propolis administered in chewing gum as compared to that incorporated in mouthwash on plaque accumulation, microbial population and patient acceptance.

DETAILED DESCRIPTION:
The study is a two parallel arms randomized controlled clinical trial where 60 high caries risk children of 6-8 years will be selected from outpatient clinic of Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Alexandria University, after securing the necessary consents. The children will be divided randomly into two equal groups (30 children each).

ELIGIBILITY:
Inclusion Criteria:

* Patients with high caries risk; who have any one of the following condition: visible cavities or radiographic penetration into the dentin, white spots on smooth surfaces, restorations within last three years due to caries.
* Free of any systemic condition.
* Cooperative children according to Frankl rating scale including positive and definitely positive scores.
* Parental acceptance

Exclusion Criteria:

* Previous use of any propolis containing products.
* Received any antibiotic 2 weeks before or during the study.
* Oral infection that compromises the mastication process.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2019-02-10 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Change in Plaque Accumulation | Baseline and after 2 weeks
  All children will be examined clinically using the Plaque Control record (O' Leary, Darke and Naylor).
  The child will be asked to chew a disclosing tablet and let it mix with saliva for 30 seconds and spit it out.
  Each tooth is divided into 4 surfaces; the plaque accumulations on all surfaces will be scored.
  The number of positively scored units is divided by the total number of tooth surfaces evaluated, and the result is multiplied by 100 to express the index as a percentage.
Microbiological Sampling of Dental Plaque | Baseline and after 2 weeks
  On the day of sampling, each child will refrain from tooth brushing in the morning, eating or drinking (except water) at least two hours before sampling time. The plaque will be collected using sterilized toothpicks. Two plaque samples will be collected from each child. Anteriorly, this will be gathered from the buccal and palatal surface of the upper incisors and canines. While posteriorly, the plaque sample will be collected from the upper and lower molars. Finally, each plaque sample will be inoculated in separate vials; each vial contains 1 ml sterile brain heart infusion broth and will be sent to the lab. After 14 days, another plaque sample will be collected as previously mentioned.
Assessment of Patient's Acceptance | After 2 weeks of treatment
  Using Visual Analogue Scale (VAS).Each patient will receive the scale form and instructed to place a vertical mark according his or her personal rating of the preparation received during the treatment period on a horizontal line scaled from 0 to 10 where 0 presented for unacceptable and 10 for acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Hend S El-Allaky, Principal Investigator — Alexandria University; Nadia A Wahba, Study Director — Alexandria University; Dalia AM Talaat, Study Director — Alexandria University; Azza S Zakaria, Study Director — Faculty of Pharmacy, Alexandria University
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Imfeld T. Chewing gum--facts and fiction: a review of gum-chewing and oral health. Crit Rev Oral Biol Med. 1999;10(3):405-19. doi: 10.1177/10454411990100030901. PMID 10759416
- [Background] Balouiri M, Sadiki M, Ibnsouda SK. Methods for in vitro evaluating antimicrobial activity: A review. J Pharm Anal. 2016 Apr;6(2):71-79. doi: 10.1016/j.jpha.2015.11.005. Epub 2015 Dec 2. PMID 29403965
- [Background] Santos FA, Bastos EM, Maia AB, Uzeda M, Carvalho MA, Farias LM, Moreira ES. Brazilian propolis: physicochemical properties, plant origin and antibacterial activity on periodontopathogens. Phytother Res. 2003 Mar;17(3):285-9. doi: 10.1002/ptr.1117. PMID 12672164
- [Background] Dodwad V, Kukreja BJ. Propolis mouthwash: A new beginning. J Indian Soc Periodontol. 2011 Apr;15(2):121-5. doi: 10.4103/0972-124X.84379. PMID 21976834